CLINICAL TRIAL: NCT00611364
Title: Physical Therapy for Hipertensive Elderly: Effects in the Physical Activity and Exercise Adherence
Brief Title: Physical Therapy for Hypertensive Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Liga de Hipertensão Arterial da Universidade Federal de Goiás (Unknown)
Responsible Party: Paulo César Brandão Veiga Jardim, Liga de Hipertensão Arterial da Universidade Federal de Goiás
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Vitorino; 0136/03
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-01

CONDITIONS: Hypertension
Keywords: Physical therapy; hypertension; aged; exercise; Physical exercise; Physical activity
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental)
  Interventions: Other: Physical Therapy and education meetings
- Control group (Active Comparator)
  Interventions: Other: education meetings

INTERVENTIONS:
Other: Physical Therapy and education meetings — Physical therapy was realized three two times per week and education meeting every fifteen days
  Arms: Study group
Other: education meetings — This group only participed of education meeting (every fifteen days)
  Arms: Control group

SUMMARY:
Physical therapy for hipertensive elderly: effects in the physical activity and exercise adherence.

Introduction: The arterial hypertension (AH) is a clinical syndrome characterized by blood pressure ≥ 140/90mmHg. Practical of physical activity (PA) and/or physical exercise (PE) is one of the modalities of not farmacological treatment. Hypertensive aged not adhere to this recommendation for presenting factors that make it difficult this practical. Objective: to verify if physical therapy (PT) treatment can improve the AF and EF adhesion of hypertensive aged. Methods: The sample was composed by 43 hypertensive aged of Arterial Hypertensive League of the Federal University of Goiás. Of these, 30 had remained in the study and had been randomized in study group (SG) (16 patients) and control group (CG) (14 patients). SG was submitted of the PT treatment and participated of educative meetings, the CG only participated of the meetings. To evaluate adhesion to the AF was used the pedometer and EF was used a questionnaire of open and closed questions, six minute walk test (6'WT) and ergometric test (ET).

ELIGIBILITY:
Inclusion Criteria:

* age or over 60 years,
* both sexes,
* regular frequency of hypertension league;
* practice of physical exercise irregular or absent (reported by professionals objectively on the record)and signature of informed consent. -

Exclusion Criteria:

* participate in another research project;
* refuse to sign the informed consent.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-03; Primary Completion 2004-09 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
to verify if physical therapy (PT) treatment can improve the AF and EF adhesion of hypertensive aged | nine months

SECONDARY OUTCOMES:
To evaluate adhesion to the AF was used the pedometer and EF was used a questionnaire of open and closed questions, six minute walk test (6'WT) and ergometric test (ET) | Nine months

CONTACTS AND LOCATIONS:
Overall Officials: Priscila Vitorino, MsD, Principal Investigator — Liga de Hipertensão Arterial da Universidade Federal de Goiás; Paulo César Jardim, PhD, Study Chair — Liga de Hipertensão Arterial da Universidade Federal de Goiás; Flávia Nogueira, Specialist, Study Chair — Liga de Hipertensão Arterial da Universidade Federal de Goiás; Juliana Brandão, Specialist, Study Chair — Liga de Hipertensão Arterial da Universidade Federal de Goiás; Haden Lobo, Specialist, Study Chair — Liga de Hipertensão Arterial da Universidade Federal de Goiás
Locations (1):
- Liga de Hipertensão Arterial da Universidade Federal de Goiás, Goiânia, Goiás, Brazil